CLINICAL TRIAL: NCT04373070
Title: CAir: Quality-of-Life Management for COPD Patients
Brief Title: Quality-of-Life Management for COPD Patients
Acronym: CAir
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Zurich (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 2020-00707
Record Dates: First submitted 2020-04-24; First posted 2020-05-04 (Actual); Last update posted 2022-11-08 (Actual); Status verified 2022-11

CONDITIONS: Copd; Chronic Respiratory Disease
Keywords: telemonitoring; chatbot; multimodal intervention
MeSH Terms: conditions — Pulmonary Disease, Chronic Obstructive | interventions — carboxyaminoimidazole ribotide

STUDY DESIGN:
Intervention Model Description: We will perform a 2:1 randomised, two-arm, single (assessor)-blind, monocentric trial.
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- chatbot-based intervention programme (intervention) (Experimental): Participants randomised to the intervention group will receive a CAir desk and a chatbot-based intervention programme for a period of 12 weeks. The CAir desk is supplied to assess HrQoL, physical activity, and spirometry data. The first week is equal to the procedure in the control group (for details see paragraph below) and serves for baseline measurements of daily physical activity. Starting in week 2 of the study duration, participants receive feedback on their daily physical activity through the CAir chatbot application and aim to increase their daily step count by 15% from baseline. Furthermore, the CAir chatbot provides several components of the "Living well with COPD" programme (e.g. educational content, information on exercise training) to the patient.
  Interventions: Combination Product: CAir
- Usual care group (control) (Other): Participants randomised to the control group receive usual care and a CAir desk for a period of 12 weeks. The CAir desk is supplied to assess daily symptom burden, physical activity, and spirometry data. In contrast to the intervention group, participants do not receive feedback or scores of the daily reported CAT and daily physical activity.
  Interventions: Combination Product: CAir

INTERVENTIONS:
Combination Product: CAir — The CAir desk is a custom-built home disease monitoring device. The device consists of a smartphone (A320 [2017], Samsung Group, Seoul, Korea), home spirometer (Air Next Spirometer, NuvoAir, Stockholm, Sweden), physical activity tracker (Charge 3, Fitbit Inc., San Francisco CA, USA), and an air-quality monitor (Foobot, Airboxlab, Esch sur Alzette, Luxembourg). The components of the CAir desk are CE-certified.

SUMMARY:
The investigators aim to investigate the effects of a telemonitoring and chatbot-based application of "Living well with COPD" (CAir) on health-related quality-of-life in patients with COPD.

DETAILED DESCRIPTION:
The disease management programme "Living well with COPD" was developed to relieve symptoms and prevent exacerbations. It covers a disease self-management approach, educational topics, lifestyle coaching and physical activity advice.

Future implications should aim to make the intervention easily accessible for a broad spectrum of patients at scalable costs. Patients need an engaging communication platform which can inform, coach and even listen in between medical visits. The inclusion of a chatbot agent may provide this tailored feedback. The investogator's aim is to investigate the effects of a telemonitoring and chatbot-based application of "Living well with COPD" on health-related quality-of-life in patients with COPD.

ELIGIBILITY:
Inclusion Criteria:

• Diagnosed COPD according to GOLD-guidelines

Exclusion Criteria:

* Physical or intellectual impairment precluding informed consent or protocol adherence
* Non-German speaking
* Acute or recent (within the last 6 weeks) exacerbation of COPD
* Attending a pulmonary rehabilitation program within the last 3 months
* Pregnant patients

Min Age: 40 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 35 (Actual)
Dates: Start 2021-02-03 (Actual); Primary Completion 2022-05-30 (Actual); Study Completion 2022-05-30 (Actual)

PRIMARY OUTCOMES:
Health-related quality-of-life (HrQoL) | 3 months
  St. George Respiratory Questionnaire (SGRQ). Scoring: Scores range from 0 to 100, with higher scores indicating more limitations.

SECONDARY OUTCOMES:
Symptom burden | 3 months
  COPD Assessment Test (CAT). Scoring: Scores range from 0-40, with higher scores indicating more symptoms.
Spirometry | 3 months
  Forced expiratory volume in one second (FEV1) in liters and percent predicted.
Spirometry | 3 months
  Forced vital capacity (FVC) in liters and percent predicted.
Accelerometry | 3 months
  Daily step count (number of steps)
Functional exercise capacity | 3 months
  Six-minute walk test (6MWT) in meters walked.
Functional exercise capacity | 3 months
  One-minute sit-to-stand test (1MSTS) in repetitions performed.

CONTACTS AND LOCATIONS:
Overall Officials: Christian F Clarenbach, MD, Principal Investigator — University of Zurich
Locations (1):
- University Hospital Zurich, Zurich, Switzerland

IPD SHARING:
Plan to Share IPD: Yes
upon reasonable request
Supporting Information: Study Protocol, SAP, ICF, CSR, Analytic Code

REFERENCES:
- [Derived] Gross C, Kohlbrenner D, Clarenbach CF, Ivankay A, Brunschwiler T, Nordmann Y, V Wangenheim F. A Telemonitoring and Hybrid Virtual Coaching Solution "CAir" for Patients with Chronic Obstructive Pulmonary Disease: Protocol for a Randomized Controlled Trial. JMIR Res Protoc. 2020 Oct 22;9(10):e20412. doi: 10.2196/20412. PMID 33090112